CLINICAL TRIAL: NCT02978846
Title: Patient Perceptions of Side Effects of Cancer Chemoradiotherapy
Brief Title: Perceptions of Side Effects of Cancer Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-15-17; NCI-2016-01260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-15-17 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-12-01 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Malignant Neoplasm; Side Effect
MeSH Terms: conditions — Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (side effects evaluation using cards): Patients are shown two groups of cards on the last day of radiation treatment. Group A lists 48 physical side effects and group B lists 27 psychosocial side effects. The cards are shuffled and patients view one card at a time and select the side effects they attribute to their current treatment. Patients rank the selected cards from each group by order of severity. The top 5 cards from each group are then shuffled together and patients rank the remaining 10 cards in order of severity.
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — Undergo side effects evaluation using cards

SUMMARY:
This study is asking patients who are undergoing radiation therapy with or without chemotherapy on how well they evaluate their side effects on the last day of treatment. This study is not to change health outcomes of the patients in this study. Asking patients to rank side effects in order of which ones bother them the most may help researchers identify the most troubling side effects of cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the perceptions of side effects and their subjective severity of patients treated with radiotherapy with and without concurrent chemotherapy at Los Angeles County (LAC) + University of Southern California (USC) Medical Center.

SECONDARY OBJECTIVES:

I. To identify the most troubling side effects of patients treated with radiotherapy with and without concurrent chemotherapy at LAC+USC Medical Center.

II. To evaluate the impact of chemotherapy combined with radiation therapy, in regards to whether or not perceptions of side effects are altered by what cancer treatment is given.

OUTLINE:

Patients are shown two groups of cards on the last day of radiation treatment. Group A lists 48 physical side effects and group B lists 27 psychosocial side effects. The cards are shuffled and patients view one card at a time and select the side effects they attribute to their current treatment. Patients rank the selected cards from each group by order of severity. The top 5 cards from each group are then shuffled together and patients rank the remaining 10 cards in order of severity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Has received at least 4 consecutive weeks of definitive radiation treatment, with or without concurrent chemotherapy
* Has not received greater than 4 weeks of chemotherapy prior to radiation therapy start
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients with either a central nervous system (CNS)-primary cancer or with brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients undergoing radiation therapy with or without chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Identify the most common type of side effects as perceived by patients on the last day of radiation treatment | Up to 1 year
  Tables and bar charts will be used to display the 10-20 highest ranked side effects overall, by sex and concurrent chemotherapy. Descriptive statistics such as means and standard deviation will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Williams, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Williams PA, Cao S, Yang D, Jennelle RL. Patient-reported outcomes of the relative severity of side effects from cancer radiotherapy. Support Care Cancer. 2020 Jan;28(1):309-316. doi: 10.1007/s00520-019-04820-2. Epub 2019 May 2. PMID 31044307